CLINICAL TRIAL: NCT06027957
Title: Phase I Clinical Trial Evaluating the Safety and Efficacy of Point-of-care CAR-T-cell Therapy in the Treatment of Relapsed/Refractory CD19+ Non-Hodgkin Lymphoma and Acute Lymphoblastic Leukemia
Brief Title: CD19 CAR T-Cell Therapy for R/R Non-Hodgkin Lymphoma and Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Collaborators: National Institute of Hematology and Blood Transfusion, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC19.26
Record Dates: First submitted 2023-07-28; First posted 2023-09-07 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: B-Cell Non Hodgkin Lymphoma; B-Cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Regimen (Experimental): * Experimental: Treatment Regimen.
  * Leukapheresis to collect white blood cells using Spectra Optia Apheresis system.
  * T cells selection, transduction, and CAR T-cell manufacturing using CliniMACS Prodigy. During this process, T cells will be genetically modified to express CD19 CAR.
  * Lymphodepleting chemotherapy conditioning regimen for 3 days.
  * CAR T-cells targeting CD19 will be infused intravenously at a dose between 1 and 2x10e6 cells/kg for 15-30 minutes.
  * Following the T-cell infusion, patients will stay in the clinic for approximately 21-28 days to monitor toxicity.
  * Outpatient follow-up will take place after 1 month, 3 months, and 6 months after infusion.
  Interventions: Biological: anti-CD19 CAR T-cells

INTERVENTIONS:
Biological: anti-CD19 CAR T-cells — For Biological: CD19 CAR T-cells
  * Dose: 1-2.10e6 cells/kg of weight
  * Route: intravenous infusion
  For Chemotherapy Drug:
  * Fludarabine (30 mg/m2/day) given intravenously (IV) on day -5 to -3.
  * Cyclophosphamide 500 mg/m2/day for NHL and 250 mg/m2/day for ALL given IV from day -5 to -3.
  * Mesna 500 mg/m2/day for NHL and 250 mg/m2/day for ALL, divided in three infusions: one day before the cyclophosphamide infusion, and 4 and 8 hours after.
  Other Names: Chemotherapy Drug

SUMMARY:
* Brief Summary: Cluster of differentiation 19 (CD19) is expressed on B cells. CD19+ tumor cells in patients with non-Hodgkin lymphoma and acute lymphoblastic leukemia can be targeted using T cells expressing CD19-specific chimeric antigen receptor (CAR).
* Objective: This study aims to evaluate the safety and efficacy of single-dose anti-CD19 CAR T-cell therapy in the treatment of relapsed/refractory CD19+ non-Hodgkin lymphoma and acute lymphoblastic leukemia.
* Eligibility: People aged 1 to 60 years with relapsed/refractory CD19+ non-Hodgkin lymphoma and acute lymphoblastic leukemia.
* Design: Phase 1 clinical trial, uncontrolled, single dose of CD19 CAR T-cells.

DETAILED DESCRIPTION:
Objectives:

* Evaluate the frequency and severity of adverse events and serious adverse events (AEs/SAEs) of the therapy.
* Evaluate the response rate after CD19 CAR T-cell infusion according to the following criteria:

  * Proportion of patients with complete response and partial response after CD19 CAR T-cell infusion
  * Progression-free survival (PFS) after infusion of CD19 CAR T-cells
  * Event-free survival (EFS) after infusion of CD19 CAR T-cells
  * Overall survival (OS) after infusion of CD19 CAR T-cells

ELIGIBILITY:
Inclusion criteria:

* B-cell acute lymphoblastic leukemia: refractory to two cycles of chemotherapy, relapsed after chemotherapy, or hematopoietic stem cell transplantation.
* B-cell non-Hodgkin lymphoma: refractory to two lines of chemotherapy, relapsed after chemotherapy, or hematopoietic stem cell transplantation.
* Age: From 1 to 60 years old (both males and females)
* Adequate organ functions:

  * Serum creatinine ≤ 1.5 x ULN or eGFR ≥ 60 mL/min/1.73 m2
  * ALT and AST ≤ 5 x ULN; Bilirubin ≤ 2.0 mg/dl
  * No chronic lung diseases, such as obstructive pulmonary disease or bronchial asthma, required continuous medications without respiratory failure (SpO2 oxygen saturation > 92% at room temperature).
  * No arrhythmia, no intracardiac thrombus or vascular wall, no heart failure, LVEF ≥ 45%
* Blood test:

  * Absolute neutrophil count (ANC) ≥ 1,000/mm3 (1 G/l) without filgrastim
  * Absolute lymphocyte count ≥ 100/mm3 (0.1 G/l)
  * Absolute platelet count ≥ 75,000/mm3 (75 G/l)
  * Hemoglobin ≥ 8.0 g/dl
* Positive for CD19 measured by immunohistochemistry or flow cytometry.
* Agree to participate in the study
* Agree to use safe methods of contraception for female patients.

Exclusion criteria:

* Involved central nervous system invasion at the time of screening.
* Medical history of veno-occlusive disease (VOD).
* Required acute treatment due to tumors such as intestinal obstructions, vascular compression, or respiratory failure.
* Having active hemolytic anemia.
* Diagnosed with primary immunodeficiency.
* Medical history of autoimmune neurological diseases or neuromyelitis.
* Receiving immunosuppressive medication, except for ≤ 30 mg prednisolone or equivalent at the time of CAR-T-cell transfusion.
* Having acute, progressive, or chronic graft-versus-host disease (GvHD).
* Having active infectious diseases determined by clinical, imaging, or other laboratory tests (blood culture, PCR, etc.)
* Patients who are critically ill or at risk of premature death characterized by:

  * Acute liver failure requiring dialysis
  * Heart failure requiring vasopressors
  * Systemic infection unresponsive to antibiotics
  * ECOG performance status ≥ 3 points at the time of screening
* Having other severe concomitant diseases (e.g., uncontrolled arterial hypertension, heart failure NYHA III-IV).
* Unstable angina within 3 months prior to screening.
* Any previous or concurrent malignancy was not B-cell lymphoma or B-ALL.
* Medical history of clinically relevant central nervous system disease, such as epilepsy, convulsions, paralysis, aphasia, uncontrolled cerebrovascular disease, traumatic brain injury, and Parkinson's disease.
* Intolerance to excipients from cellular products.
* Pregnant women or those who expect to be pregnant or reastfeeding.
* Other diseases or other conditions and circumstances that, according to the investigator's assessment, make it difficult to ensure compliance with study treatment.
* Participation in another clinical trial at the time of screening

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the frequency and severity of adverse events and serious adverse events (AEs/SAEs) of the therapy | 6 months
  The incidence of adverse events (AEs) and serious adverse events (SAEs) will be recorded and classified according to CTCAE v5 (grade 1-5). CRS and ICANs will be classified using the ASTCT criteria (grade 1-5). These parameters will be used to assess the safety of the therapy.

SECONDARY OUTCOMES:
Proportion of patients with complete response and partial response after CD19 CAR T-cell infusion (%) | Day 30 and day 90 after CAR-T infusion for B-ALL; day 90 after CAR-T infusion for NHL
  Patients with B-ALL will receive bone marrow biopsy assessed on day 30 and day 90 to check blast frequency and MRD. The response will be classified according to NCCN guidelines.
  Patients with NHL will be examined PET-CT or CT on day 90. The response will be classified according to Cheson guidelines.
Progression-free survival (PFS) (months) | 6 months
  PFS is defined as the time from CAR T-cell infusion, until disease progression or death from any cause. Progression is defined as an increase of tumor load, the development of new lesions.
Event-free survival (EFS) (months) | 6 months
  EFS is defined as time to treatment failure (including complete remission with incomplete hematologic or platelet recovery), relapse from complete remission, or death from any cause.
Overall survival (OS) (months) | 6 months
  EFS is defined as time to death

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Liem Nguyen, PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No